CLINICAL TRIAL: NCT06151262
Title: A Single-arm, Exploratory Clinical Study of Trilaciclib Combined With mFOLFIRINOX Regimen in the Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: A Study of Trilaciclib Combined With mFOLFIRINOX in the Treatment of Patients With Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-419-02
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib+mFOLFIRINOX (Experimental): The treatment regimen was as follows:
  Trilaciclib 240mg/m2 IV infusion, D1, D2，Q2W； Oxaliplatin 68mg/m2 IV infusion, D1; Irinotecan 135mg/m2 IV infusion D1; leucovorin 400mg/m2 IV infusion D1; 5-FU 2.4g/m2 IV infusion for 46h, D1; A total of 12 cycles of treatment were performed every 14 days as a cycle.
  Interventions: Drug: Trilaciclib+mFOLFIRINOX

INTERVENTIONS:
Drug: Trilaciclib+mFOLFIRINOX — This was a single-arm, exploratory study of the combination of Trilaciclib and mFOLFIRINOX in patients with advanced pancreatic cancer receiving first-line therapy. Observed the incidence of chemotherapy-induced myelosuppression, and imaging was performed every four cycles to assess tumor response.
  Other Names: G1T28; CDK 4/6 inhibitor

SUMMARY:
To observe the incidence of chemotherapy-induced myelosuppression and the safety of Trilaciclib combined with mFOLFIRINOX in patients with advanced pancreatic cancer receiving first-line treatment.

DETAILED DESCRIPTION:
This study was a single-arm, exploratory clinical study. Patients with advanced pancreatic cancer were screened and enrolled according to the inclusion and exclusion criteria described in the study protocol. Informed consent was signed after full communication. Patients with advanced pancreatic cancer who received first-line treatment were treated with Trilaciclib +mFOLFIRINOX. The incidence of chemotherapy-induced myelosuppression was used as the primary endpoint to observe whether Trilaciclib could reduce the occurrence or degree of chemotherapy-induced myelosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* ECOG score 0 or 1
* Expected survival≥12 weeks
* Patients with histologically or cytologically confirmed pancreatic cancer
* Have not received any antineoplastic therapy prior to treatment
* Major organ functions within 7 days prior to treatment shall meet the following criteria: a. Neutrophil count ≥1.5×109 /L； b. Hemoglobin ≥10g/dL； c. Platelet count ≥100×109 /L
* Biochemical examination shall meet the following standards: a、Total bilirubin(TBIL)≤1.5times the upper limit of normal value(ULN); b、ALT and AST≤1.5×ULN ; c、creatinine clearance(CCr)≥60ml/min
* Patients of reproductive age(including female and male patients'female companions)must use effective birth control measures
* Subjects voluntarily joined the study and signed an informed consent form(ICF)
* It is expected that the patient has good compliance and can follow up the efficacy and adverse reactions according to the protocol requirements

Exclusion Criteria:

* Had received systemic antineoplastic therapy
* Pregnant and lactating women. Women of childbearing age had to test a negative pregnancy test within 7 days before enrollment
* Substance abuse, clinical or psychological or social factors that may interfere with informed consent or the conduct of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of CIM | During treatment. Treatment cycles of 14 days continued from the first dose until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator (up to 24 months）
  Incidence of chemotherapy-induced myelosuppression

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death(up to 24 months)
  Overall survival defined as time from the date of first dose of study drug to death due to any cause for those who died; or time to last contact known as alive for those who survived in the study (censored cases)
PFS | From date of first dose of study drug to radiographic disease progression（Up to 24 months）
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurs first.
Safety and Tolerability | Up to 36 months
  Occurrence and severity of AEs by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: du juan, M.D., Principal Investigator — The Affiliated Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No